CLINICAL TRIAL: NCT03952351
Title: Troponin in Acute Chest Pain to Risk Stratify and Guide EffecTive Use of Computed Tomography Coronary Angiography
Acronym: TARGET-CTCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); University of Sheffield (Other); NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AC18106
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTCA with standard care (Experimental): Patients will be referred for CT Coronary Angiography, ideally within 2 weeks of randomisation
  Interventions: Radiation: CT Coronary Angiography (CTCA)
- Standard care (No Intervention)

INTERVENTIONS:
Radiation: CT Coronary Angiography (CTCA) — CTCA scan in accordance with British Society of Cardiovascular Imaging CT guidelines
  Arms: CTCA with standard care

SUMMARY:
Most patients presenting to hospital with symptoms of a heart attack are sent home without further tests once a heart attack has been ruled out. Current strategies to assess patients with a suspected heart attack involve blood tests to measure troponin, a protein released into the bloodstream when the heart muscle is damaged.

Despite having had a heart attack ruled-out, some patients have unrecognised heart disease and are at risk of having a heart attack in the future. However, clinicians do not know what is the best approach to identify and treat these patients.

This study will use a heart scan known as computed tomography coronary angiogram (CTCA) to look for unrecognised heart disease in patients who have had a heart attack ruled out. In an earlier study, the Investigators performed this scan in patients referred to the outpatient cardiology clinic with stable chest pain and found that this improved the diagnosis of heart disease, leading to improvement in patient care that prevented future heart attacks.

Previous research from the Investigators has also found that troponin levels below those used to diagnose a heart attack may help to identify those who are at greater risk of having a heart attack in the future.

The aim of this study is to find out if patients with these low levels of troponin, where a heart attack has been ruled out, will benefit from CTCA to look for unrecognised coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to hospital with symptoms of suspected acute coronary syndrome
* Age 18 years and over
* Maximum high-sensitivity cardiac troponin concentration between 5ng/L and the 99th percentile

Exclusion Criteria:

* Diagnosis of myocardial infarction during index presentation
* Clear alternative diagnosis or participant requires further inpatient clinical assessment
* Recent CTCA or invasive coronary angiogram (within 1 year)
* Patient inability to undergo CT scanning, e.g. due to severe renal failure (estimated glomerular filtration rate <30 mL/min) or major allergy to iodinated contrast media
* Current pregnancy or breast feeding
* Inability to give informed consent
* Further investigation for coronary artery disease would not be in the patient's interest, e.g. due to limited life expectancy, quality of life or functional status
* Previous randomisation into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3170 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Composite of myocardial infarction or cardiac death | Randomisation through to study completion, median duration of 36 months
  The first event of myocardial infarction or cardiac death

SECONDARY OUTCOMES:
Myocardial Infarction | Randomisation through to study completion, median duration of 36 months
  The first event of myocardial infarction (MI). MI will be defined according to the 4th Universal Definition of Myocardial Infarction
Cardiac death | Randomisation through to study completion, median duration of 36 months
  Cardiac death will be defined as death resulting from an acute myocardial infarction, sudden cardiac death, or death due to heart failure.
Cardiovascular death | Randomisation through to study completion, median duration of 36 months
  Cardiovascular death will be defined as death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular haemorrhage, and death due to other cardiovascular causes
Non-cardiovascular death | Randomisation through to study completion, median duration of 36 months
All-cause death | Randomisation through to study completion, median duration of 36 months
Unscheduled urgent coronary revascularisation | Randomisation through to study completion, median duration of 36 months
  Unscheduled urgent coronary revascularisation will be identified via record linkage from central NHS registers (e.g. the Scottish Morbidity Register by the Information Services Division (ISD) Scotland) or from extracts obtained from the participating hospitals electronic patient record system.
Hospital reattendance with suspected ACS | Randomisation through to study completion, median duration of 36 months
  Reattendance with suspected ACS will be defined as any unscheduled hospital attendance where cardiac troponin testing is performed for suspected ACS following randomisation
Proportion of patients with major bleeding (BARC 3-5) | Randomisation through to study completion, median duration of 36 months
  Bleeding will be defined according to the Bleeding Academic Research Consortium (BARC) definition of bleeding. We will use pre-defined codes from International Classification of Diseases (ICD-10) and Office of Population Censuses and Surveys (OPCS) to classify each bleeding event as per the BARC definition.
Symptomatic status as assessed by the short form Seattle Angina Questionnaire (SAQ-7) | 3, 12 and 24 months
Quality of life as assessed by the EQ-5D-5L | 3, 12 and 24 months

OTHER OUTCOMES:
Proportion of patients with allergy/anaphylaxis/acute kidney injury following study CTCA scan | 2 weeks
Proportion of patients undergoing non-study CTCA or invasive coronary angiography (ICA) | 90 days
Proportion of patients with clinically significant abnormal non-cardiac findings on study CTCA scan | 2 weeks
Dose length product from study CTCA scan | 2 weeks
Proportion of patients undergoing non-invasive stress test (cost-effectiveness) | 90 days
Proportion of patients prescribed therapies for coronary artery disease (cost-effectiveness) | Randomisation through to study completion, median duration of 36 months
Proportion of patients undergoing planned revascularisation (cost-effectiveness) | Randomisation through to study completion, median duration of 36 months
Incremental cost per quality-adjusted life year (QALY) gained (cost-effectiveness) | Randomisation through to study completion, median duration of 36 months

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - Lewisham & Greenwich NHS Trust, London
  - Milton Keynes University NHS Hospital, Milton Keynes
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - University Hospital Southampton NHS Trust, Southampton
  - North Tees NHS Hospital Foundation, Stockton
  - Torbay & South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the primary paper, a deidentified individual participant data set will be will be made available for data sharing purposes, subject to necessary governance approvals. Access to the deidentified dataset will be under a controlled access model.

REFERENCES:
- [Derived] Lee KK, Lowe D, O'Brien R, Wereski R, Bularga A, Taggart C, Lowry MTH, Ferry AV, Williams MC, Roditi G, Byrne J, Tuck C, Cranley D, Thokala P, Goodacre S, Keerie C, Norrie J, Newby DE, Gray AJ, Mills NL. Troponin in acute chest pain to risk stratify and guide effective use of computed tomography coronary angiography (TARGET-CTCA): a randomised controlled trial. Trials. 2023 Jun 13;24(1):402. doi: 10.1186/s13063-023-07431-9. PMID 37312104